CLINICAL TRIAL: NCT03005067
Title: A Randomized, Parallel-Group, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy and Safety of 1146A Nasal Spray in Adult Subjects With Symptoms of Common Cold
Brief Title: To Evaluate the Efficacy and Safety of 1146A Nasal Spray in Adult Participants With Symptoms of Common Cold
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205684
Record Dates: First submitted 2016-12-07; First posted 2016-12-29 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — carbomer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Carbomer 980 (1146A) (Experimental): Participants will be administered test product (nasal spray) containing carbomer 980 gel. Three actuations per nostril per dose will be applied, each actuation will be 140µL (microliters) i.e. equivalent to 140mg.
  Interventions: Drug: Carbomer 980 (1146A)
- Placebo (Placebo Comparator): Participants will be administered reference product (nasal spray) containing vehicle without carbomer 980. Three actuations of placebo nasal spray per nostril per dose; each actuation will be 140µL.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Carbomer 980 (1146A) — Test product containing carbomer 980 gel
  Arms: Carbomer 980 (1146A)
Other: Placebo — Reference product containing vehicle without carbomer 980 gel
  Arms: Placebo

SUMMARY:
This study will be conducted in adult participants with symptoms of common cold assessing if 1146A nasal spray reduces the severity of symptoms of the common cold compared to placebo. The study will also evaluate the safety of 1146A compared to placebo.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, parallel-group, double blind, 2-arm, placebo controlled study to evaluate the efficacy and safety of 1146A in adult participants with symptomatic common cold in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 to 75 years inclusive.
* Male or female.
* Good general and mental health with, in the opinion of the Investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical and Investigator-led nasal examination.
* Females of childbearing potential who are, in the opinion of the Investigator, practicing a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone OR injectable progestogen OR implants of levonorgestrel OR estrogenic vaginal ring OR percutaneous contraceptive patches OR intrauterine device or intrauterine system OR double barrier method (condom or occlusive cap (diaphragm or cervical vault caps) plus spermicidal agent (foam, gel, film, cream, suppository)) OR male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant.
* Investigator confirmed diagnosis of symptomatic common cold with an onset of less than 48 hours prior to randomization. Symptomatic common cold is defined as TSS > 9 AND a score >1 for at least one of the following symptoms: sore throat, runny nose, or blocked nose.

Exclusion Criteria:

* Women who have a positive urine pregnancy test.
* Women who are breast-feeding.
* During the entire study (Screening - last participant visit):
* A. Participant who have used medications or therapies that could interfere with study evaluations and have not had the proper washout period from these medications or therapies or are anticipated to require any concomitant intranasal medication during that period or at any time throughout the study.
* B. Nasal disease(s) likely to affect deposition of intranasal medication, such as chronic sinusitis, rhinitis medicamentosa, clinically significant polyposis, or clinically significant nasal structural abnormalities.
* C. Nasal surgery or sinus surgery within the previous year.
* D. Any condition that prohibits the participant from actuating nasal spray devices (severe rheumatoid arthritis; deformed hands and fingers; missing fingers).
* E. Clinically relevant abnormal physical findings which, in the opinion of the Investigator or sponsor's medical monitor, would interfere with the objectives of the study or that may preclude compliance with the study procedures.
* F. Uncontrolled cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrine, metabolic, autoimmune, neurological, psychiatric or other diseases at screening that would interfere with the study in the opinion of the Investigator.
* G. Participants with seasonal allergic rhinitis if randomization occurs during their expected allergy season or perennial allergic rhinitis.
* H. Severe COPD, persistent asthma, or recent COPD/asthma exacerbation.
* I. An inability to comprehend and satisfactorily use the measurement instruments as determined by the study sites staff on screening.
* J. Participants with a fever > 38°C (100.4°F).
* K. Frequent uses of analgesics (i.e. have taken an analgesic for pain in headache and pain in muscle/joints for at least 1 dose per week on average over the past 6 months).
* Known or suspected intolerance or hypersensitivity to any of the study medications, excipients or investigational device material or to medications of similar chemical classes, any history of drug hypersensitivity or other significant allergic diathesis that could affect study participation and known or suspected contraindications, including history of allergy or photosensitivity to study medication/s.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit or 5 half-lives of enrollment, whichever is longer and previous participation in this study (i.e. participants cannot be re-screened or randomized).

Recent history (within the last 5 years) of alcohol or other substance abuse and positive urine drug screen.

* An employee of the sponsor or the study sites or members of their immediate family and persons directly or indirectly involved in the execution of this protocol, including employees of the contract research organization (CRO) and persons related to them.
* On nasal examination by Investigator, the presence of nasal disease likely to affect deposition of intranasal treatment or any superficial or moderate nasal mucosal erosion, nasal mucosal ulceration, or nasal septum perforation at the screening visit. Participants with difficulty in using the nasal spray applicator, "vulnerable" individual (as defined by the IRB e.g. incarcerated person) and any condition not identified in the protocol that in the opinion of the Investigator would confound the evaluation and interpretation of the study data or may put the participant at risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (24):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Elkhorn, Nebraska
  - GSK Investigational Site, Fremont, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Vineland, New Jersey
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Hatboro, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 24 centers in United States.
Pre-assignment Details: A total of 308 participants were screened for this study, out of which137 participants were screening failure.
Groups:
- Test Product: Participants were administered test product (nasal spray) containing carbomer 980 gel (1146A).
- Placebo Nasal Spray: Participants were administered placebo nasal spray containing vehicle without carbomer 980.
Period: Overall Study
Arm/Group | Test Product | Placebo Nasal Spray
Started | 90 | 81
Completed | 80 | 74
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 4 | 3
Not completed — Other (reason not specified) | 3 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline parameters were reported for safety population. Safety population (N=168) included all randomized participants who received at least one dose of study medication.Three participants were randomized but not dosed, therefore not included in safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Placebo Nasal Spray | Total
Number analyzed (Participants) | 87 | 81 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (13.99) | 50.3 (12.60) | 50.1 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 30 | 25 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 28 | 63
  White | 51 | 53 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Nasal Symptom Score Over Days 1-4 (ANSS1-4)
Description: The nasal symptom score (NSS) was calculated as the sum score of the nasal symptoms (runny nose, blocked nose and sneezing). The participants self-assessed each individual sign/symptom which was scored using the following 4-point scale: 0 = absent symptoms (no sign/symptom evident), 1 = mild symptoms (sign/symptom clearly present, but minimal awareness; easily tolerated), 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping);score range (Min-Max): 0-9 . The average nasal symptom score (ANSS) on days 1 to 4 was calculated as the mean of the 4 daily NSS across study days 1 to 4. A lower score reflects better nasal symptoms.
Time Frame: Up to Day 4 (Day 1 to 4)
Population: Modified Intent-to-Treat(mITT) population was the primary population of analysis. The mITT (N=165) population was defined as participants who received at least one dose of study medication and have at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Product | Placebo Nasal Spray
Number analyzed (Participants) | 86 | 79
Score on a scale | 3.428 (1.4784) | 3.336 (1.6917)
Statistical Analysis 1: Comparison: Test Product vs Placebo Nasal Spray; Test type: Other; p = 0.516, ANCOVA — P-value was based on the Wald statistic Chi-Square test, from an ANCOVA model with treatment, center, and Day 1 dosing time stratification as factors and baseline NSS (Day 1 prior to the first dose) as a covariate; Mean Difference (Net) = 0.137, 95% CI 2-sided [-0.279 to 0.553] — Difference of LS mean is 1146A Formulation Nasal Spray - Placebo Nasal Spray. 95% CI is for difference of LS means

2. Secondary Outcome: Average Nasal Symptom Score Over Days 1-7 (ANSS1-7)
Description: The nasal symptom score (NSS) was calculated as the sum score of the nasal symptoms (runny nose, blocked nose and sneezing). The participants self-assessed each individual sign/symptom which was scored using the following 4-point scale: 0 = absent symptoms (no sign/symptom evident), 1 = mild symptoms (sign/symptom clearly present, but minimal awareness; easily tolerated), 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping);score range (Min-Max): 0-9 . The average nasal symptom score (ANSS) on days 1 to 7 was calculated as the mean of the 7 daily NSS across study days 1 to 7. A lower score reflects better nasal symptoms.
Time Frame: Up to Day 7 (Day 1 to 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Product | Placebo Nasal Spray
Number analyzed (Participants) | 86 | 79
Score on a scale | 2.700 (1.3142) | 2.651 (1.5455)

3. Secondary Outcome: Average Total Symptom Score Over Days 1-4 (ATSS1-4)
Description: The total symptom scores (TSS) were calculated as the sum score of the nasal symptoms (runny nose, blocked nose and sneezing) and other symptoms (headache, muscle ache, chills, sore throat and cough). The participants self-assessed each individual sign/symptom which was scored using the following 4 point scale: 0 = absent symptoms (no sign/symptom evident), 1 = mild symptoms (sign/symptom clearly present, but minimal awareness; easily tolerated), 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping);Score range (Min-Max):0-24. Average Total Symptom Score (ATSS) on days 1 to 4 were derived as the mean of all TSS across study Days 1 to 4. A lower score reflects better nasal symptoms.
Time Frame: Up to Day 4 (Day 1 to 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Product | Placebo Nasal Spray
Number analyzed (Participants) | 86 | 79
Score on a scale | 7.811 (3.1962) | 7.754 (3.4996)

4. Secondary Outcome: Average Total Symptom Score Over Days 1-7 (ATSS1-7)
Description: The total symptom scores (TSS) were calculated as the sum score of the nasal symptoms (runny nose, blocked nose and sneezing) and other symptoms (headache, muscle ache, chills, sore throat and cough). The participants self-assessed each individual sign/symptom which was scored using the following 4 point scale: 0 = absent symptoms (no sign/symptom evident), 1 = mild symptoms (sign/symptom clearly present, but minimal awareness; easily tolerated), 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping);Score range (Min-Max):0-24. Average Total Symptom Score (ATSS) on days 1 to 7 were derived as the mean of all TSS across study Days 1 to 7. A lower score reflects better nasal symptoms.
Time Frame: Up to Day 7 (Day 1 to 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Product | Placebo Nasal Spray
Number analyzed (Participants) | 86 | 79
Score on a scale | 6.171 (2.9822) | 6.195 (3.2078)

ADVERSE EVENTS:
Time Frame: Approximately 8 days
Description: All treatment emergent adverse events and serious adverse were reported.
Arm/Group | Test Product | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/81
Other Adverse Events (participants affected / at risk) | 32/87 | 34/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (N=87) | Placebo Nasal Spray (N=81)
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (N=87) | Placebo Nasal Spray (N=81)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 4
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 3 | 2
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 2
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTRANASAL HYPOAESTHESIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NASAL MUCOSAL EROSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL MUCOSAL ULCER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RHINALGIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 8 | 6
DIZZINESS (Nervous system disorders) | 2 | 0
BURNING SENSATION (Nervous system disorders) | 0 | 1
SINUS HEADACHE (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0
ADMINISTRATION SITE PAIN (General disorders) | 0 | 3
APPLICATION SITE PAIN (General disorders) | 1 | 2
CHILLS (General disorders) | 2 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0
FEELING COLD (General disorders) | 1 | 0
FEELING JITTERY (General disorders) | 0 | 1
PYREXIA (General disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 2
DRY MOUTH (Gastrointestinal disorders) | 1 | 0
RETCHING (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1
ABSCESS OF EYELID (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1
LARYNGITIS (Infections and infestations) | 0 | 1
TOOTH INFECTION (Infections and infestations) | 0 | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 | 0
BACK INJURY (Injury, poisoning and procedural complications) | 1 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 1 | 0
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 0 | 1
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 1
PRODUCT TASTE ABNORMAL (Product Issues) | 0 | 1
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03005067/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT03005067/SAP_001.pdf